CLINICAL TRIAL: NCT04980820
Title: Changes in Capillary pCO2 While Wearing FFP2 and FFP3 Masks Masks by Medical Staff - a Prospective Cross-over Study
Brief Title: Changes in Capillary Carbon Dioxide Partial Pressure (pCO2) While Wearing FFP2 / FFP3 Masks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, David M Baron, MD, Assoc. Prof. PD Dr. David Baron, EDIC, Medical University of Vienna
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 1144/2021
Record Dates: First submitted 2021-07-14; First posted 2021-07-28 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Hypercapnia
MeSH Terms: conditions — Hypercapnia

STUDY DESIGN:
Intervention Model Description: 1. arm: starts with no mask - FFP2 mask - FFP3 mask
  2. arm: starts with no mask - FFP3 mask - FFP2 mask
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FFP2 (Experimental): This arm starts with a FFP2 mask and switches to a FFP3 mask.
  Interventions: Other: No mask; Device: Filtering face mask 2 (FFP2); Device: Filtering face mask 3 (FFP3)
- FFP3 (Experimental): This arm starts with a FFP3 mask and switches to a FFP2 mask.
  Interventions: Other: No mask; Device: Filtering face mask 2 (FFP2); Device: Filtering face mask 3 (FFP3)

INTERVENTIONS:
Other: No mask — The participant is asked to wear no mask for 10 minutes.
Device: Filtering face mask 2 (FFP2) — The participant is asked to wear a FFP2 mask for 1 hour during work.
Device: Filtering face mask 3 (FFP3) — The participant is asked to wear a FFP3 mask for 1 hour during work.

SUMMARY:
The aim of this study is to determine whether there are any changes in the carbon dioxide partial pressure in medical staff while wearing a filtering face piece (FFP) 2 or FFP3 mask.

Furthermore, changes in the capillary oxygen partial pressure, the subjective respiratory effort and the breathing rate are measured.

DETAILED DESCRIPTION:
In the fight against the severe acute respiratory syndrome coronavirus type 2 (SARS-CoV-2), the personal protective equipment (PPE) of medical staff plays a special role. Since the pathogen can be transmitted via droplets, particle-filtering half masks (filtering face piece - FFP) are a substantial part of the PPE. The current data indicate that there may be an increase in the carbon dioxide partial pressure (PcCO2) in the blood when wearing an FFP2 / 3 mask during routine medical activity.

The aim of this prospective cross-over study is to compare the PcCO2 measured by capillary blood sampling from medical staff while wearing an FFP2 or FFP3 mask. The PcCO2 determined without a mask serves as a reference value. While no mask is worn, the PcCO2, the subjective respiratory effort, the breathing rate and the capillary oxygen partial pressure (PcO2) is measured. The study participants then wear an FFP2 or FFP3 mask for one hour, and the same parameters are collected. Subsequently, the participant switches to an FFP3 or FFP2 mask, and the last measurement is conducted after one hour.

ELIGIBILITY:
Inclusion Criteria:

* medical staff working at the Vienna General Hospital
* oral and written consent to take part voluntarily in this trial

Exclusion Criteria:

* hypersensitivity / allergy against Nonylvanillamid, Nikotinsäure-beta-butoxyethylester or other component of "Finalgon Salbe"
* not Coronavirus disease-19 vaccinated
* pregnancy
* breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change of PcCO2 | 1. measurement after 10 minutes without mask, 2. measurement after 1 hour with mask (FFP2/3), 3. measurement after 1 hour with mask (FFP3/2)
  Change of capillary carbon dioxide partial pressure (PcCO2)

SECONDARY OUTCOMES:
Change of PcO2 | 1. measurement after 10 minutes without mask, 2. measurement after 1 hour with mask (FFP2/3), 3. measurement after 1 hour with mask (FFP3/2)
  Change of capillary oxygen partial pressure (PcO2)
Respiratory rate | 1. measurement after 10 minutes without mask, 2. measurement after 1 hour with mask (FFP2/3), 3. measurement after 1 hour with mask (FFP3/2)
  Number of breaths per minute
Exertion score | 1. measurement after 10 minutes without mask, 2. measurement after 1 hour with mask (FFP2/3), 3. measurement after 1 hour with mask (FFP3/2)
  Participant subjective score: "How difficult is it for you to breathe at the moment?"; scale from 1-5, 1= easy, 2= rather easy, 3= moderate, 4= rather hard, 5= hard

CONTACTS AND LOCATIONS:
Overall Officials: Georg Röder, M.D., Principal Investigator — Medical University of Vienna, Dept. of Anaesthesiology, Critical Care and Pain Medicine
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paules CI, Marston HD, Fauci AS. Coronavirus Infections-More Than Just the Common Cold. JAMA. 2020 Feb 25;323(8):707-708. doi: 10.1001/jama.2020.0757. No abstract available. PMID 31971553
- [Background] Fletcher SJ, Clark M, Stanley PJ. Carbon dioxide re-breathing with close fitting face respirator masks. Anaesthesia. 2006 Sep;61(9):910. doi: 10.1111/j.1365-2044.2006.04767.x. No abstract available. PMID 16922771
- [Background] Ozdemir L, Azizoglu M, Yapici D. Respirators used by healthcare workers due to the COVID-19 outbreak increase end-tidal carbon dioxide and fractional inspired carbon dioxide pressure. J Clin Anesth. 2020 Nov;66:109901. doi: 10.1016/j.jclinane.2020.109901. Epub 2020 May 22. PMID 32473501
- [Background] Kim JH, Benson SM, Roberge RJ. Pulmonary and heart rate responses to wearing N95 filtering facepiece respirators. Am J Infect Control. 2013 Jan;41(1):24-7. doi: 10.1016/j.ajic.2012.02.037. Epub 2012 Sep 1. PMID 22944510
- See also: Rational use of personal protective equipment for coronavirus disease (COVID-19) and considerations during severe shortages — https://www.who.int/publications/i/item/rational-use-of-personal-protective-equipment-for-coronavirus-disease-(covid-19)-and-considerations-during-severe-shortages